CLINICAL TRIAL: NCT00053768
Title: Randomised Trial Comparing Chemotherapy Mit CHOEP (Cyclophosphamid, Doxorubicin, Vincristin, Etoposid Und Prednison) In 21-Day Intervals In Standard And Escalated Doses In Patients Aged 18-60 Years Of Age With Aggresive Non-Hodgkin-Lymphomas Favourable Prognoses
Brief Title: Combination Chemotherapy Followed By Radiation Therapy in Treating Patients With Aggressive Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: German High-Grade Non-Hodgkin's Lymphoma Study Group (Other)
Responsible Party: Sponsor
Organization: Universität des Saarlandes (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000269371; DSHNHL-1999-2; EU-20242
Record Dates: First submitted 2003-02-05; First posted 2003-02-06 (Estimated); Last update posted 2021-05-18 (Actual); Status verified 2021-05

CONDITIONS: Lymphoma
Keywords: contiguous stage II grade 3 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; stage I grade 3 follicular lymphoma; stage III grade 3 follicular lymphoma; stage IV grade 3 follicular lymphoma; contiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; stage I adult diffuse mixed cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage IV adult diffuse mixed cell lymphoma; contiguous stage II adult diffuse large cell lymphoma; contiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult Burkitt lymphoma; stage I adult diffuse large cell lymphoma; stage I adult Burkitt lymphoma; stage III adult diffuse large cell lymphoma; stage III adult Burkitt lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult Burkitt lymphoma; contiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; stage I adult immunoblastic large cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; contiguous stage II adult lymphoblastic lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; stage I adult lymphoblastic lymphoma; stage III adult lymphoblastic lymphoma; stage IV adult lymphoblastic lymphoma; contiguous stage II mantle cell lymphoma; noncontiguous stage II mantle cell lymphoma; stage I mantle cell lymphoma; stage III mantle cell lymphoma; stage IV mantle cell lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Burkitt Lymphoma; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Mantle-Cell | interventions — Filgrastim; EPOCH protocol; Cyclophosphamide; Doxorubicin; Etoposide; Prednisone; Vincristine; Radiotherapy

ARMS (2):
- CHOEP-21 (Active Comparator): CHOEP-21-Schema:
  Cyclophosphamid (750 mg/m2 i.v. d1), Doxorubicin (50 mg/m2 i.v. d1), Vincristin (2 mg i.v. d1), Etoposid (100 mg/m² i.v. d1-3), Prednison (100 mg p.o. d1-5)
  Interventions: Biological: filgrastim; Drug: EPOCH regimen; Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: etoposide; Drug: prednisone; Drug: vincristine sulfate; Radiation: radiation therapy
- high CHOEP-21 (Experimental): High-CHOEP-21-Schema:
  Cyclophosphamid (1400 mg/m2 i.v. d1), Doxorubicin (32,5 mg/m2 i.v. d1+2), Vincristin (2 mg i.v. d1), Etoposid (175 mg/m² i.v. d1-3), Prednison (100 mg p.o. d1-5)
  Interventions: Biological: filgrastim; Drug: EPOCH regimen; Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: etoposide; Drug: prednisone; Drug: vincristine sulfate; Radiation: radiation therapy

INTERVENTIONS:
Biological: filgrastim
Drug: EPOCH regimen
Drug: cyclophosphamide
Drug: doxorubicin hydrochloride
Drug: etoposide
Drug: prednisone
Drug: vincristine sulfate
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining more than one drug and giving the drugs in different ways may kill more cancer cells. Radiation therapy uses high-energy x-rays to damage cancer cells. It is not yet known which combination chemotherapy regimen followed by radiation therapy is more effective in treating aggressive non-Hodgkin's lymphoma.

PURPOSE: This randomized phase III trial is studying two combination chemotherapy regimens followed by radiation therapy to compare how well they work in treating patients with aggressive non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the efficacy of standard-dose vs high-dose cyclophosphamide, doxorubicin, vincristine, etoposide, and prednisone followed by radiotherapy, in terms of time to treatment failure, in patients with aggressive non-Hodgkin's lymphoma.
* Compare the acute and long-term toxic effects of these regimens in these patients.
* Compare the complete response rate, survival and tumor control, and disease-free survival in patients treated with these regimens.
* Analyze the time to relapse after radiotherapy in these patients.

OUTLINE: This is a randomized, open-label, multicenter study. Patients are stratified according to LDH levels (no greater than upper limit of normal [ULN] vs greater than ULN), initial bulky disease (yes vs no), stage (I or II vs II or IV), ECOG performance status (0 or 1 vs 2 or 3), and participating center. Patients are randomized to 1 of 2 treatment arms as follows:

* Arm I (Standard dose): Patients receive cyclophosphamide IV, doxorubicin IV, and vincristine IV on day 1; etoposide IV on days 1-3; and oral prednisone on days 1-5 (CHOEP) in standard doses.
* Arm II (Escalated dose): Patients receive high-dose CHOEP as in arm I. Patients also receive filgrastim (G-CSF) subcutaneously on days 6-12.

In both arms, treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

After completion of CHOEP chemotherapy, patients with initial bulky disease or extranodal involvement undergo radiotherapy 5 days a week for 4 weeks.

Patients who undergo radiotherapy are followed at 2 months after radiotherapy. All patients (including those who undergo radiotherapy) are followed every 3 months for 2 years and then every 6 months for 3 years.

PROJECTED ACCRUAL: A total of 389 patients were accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed aggressive non-Hodgkin's lymphoma

  * Previously untreated disease
* Favorable prognosis

  * International Prognostic Index score of 0-1
* No more than 25% marrow involvement

PATIENT CHARACTERISTICS:

Age

* 18 to 60

Performance status

* ECOG 0-3 OR
* Karnofsky 40-100%

Life expectancy

* Not specified

Hematopoietic

* Platelet count at least 100,000/mm^3
* WBC at least 2,500/mm^3

Hepatic

* No active hepatitis infection

Renal

* Not specified

Other

* HIV negative
* Not pregnant or nursing
* No relevant accompanying disease
* No other concurrent malignancy
* No contraindications to any study medications
* No prior noncompliance by patient

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* No prior radiotherapy

Surgery

* Not specified

Other

* No other concurrent participation in another treatment study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 392 (Actual)
Dates: Start 2002-04; Primary Completion 2006-12-05 (Actual); Study Completion 2006-12-05 (Actual)

PRIMARY OUTCOMES:
Time to treatment failure (TTF) at first relapse | 3 years within study and periodically after study completion
  Time to Treatment failure using the Kaplan_Meier-Method

SECONDARY OUTCOMES:
Complete response rate at first relapse | 3 years within study and periodically after study completion
  Number of complete remission (CR) and unconfirmed complete Remission (CRu)
Survival time | 3 years within study and periodically after study completion
  Time till death (whatever cause)
Tumor control | thought the treatment
  Calcution of treatment Duration using the Kaplan-Meier method
Disease-free survival | 3 years within study and periodically after study completion
  Time of disease-free survivial

CONTACTS AND LOCATIONS:
Overall Officials: Michael G.M. Pfreundschuh, MD, Study Chair — Universitaetsklinikum des Saarlandes
Locations (175):
- Germany (173):
  - Haematologisch Onkologische Praxis, Aachen
  - Klinikum St. Marien, Amberg
  - Gemeinschaftspraxis Fuer Innere Medizin, Haematologie Und Internistische Onkologie, Ansbach
  - Specialist Practice for Oncology, Aschaffenburg
  - II. Medizinische Klinik, Aschaffenburg
  - Haematologische Praxis, Augsburg
  - Hamatologische/Onkologische Gemeinschaftspraxis - Augsburg, Augsburg
  - Klinikum Augsburg, Augsburg
  - Kreiskrankenhaus Aurich, Aurich
  - Kreiskrankenhaus, Bad Hersfeld
  - Humaine - Clinic, Bad Saarow
  - Krankenhaus Hohe Warte Mediziniche Klinik, Bayreuth
  - Onkolog - Haematolog Schwerpunktpraxis, Berlin
  - Charite - Campus Charite Mitte, Berlin
  - Hospital Complex Bernburg, Bernburg
  - Krankenhaus Bietigheim, Bietigheim
  - Saint Agnes Hospital, Bocholt
  - Saint Josef Hospital, Bochum
  - Knappschaft Krankenhaus, Bochum
  - Medizinische Poliklinik, Bonn
  - Rheinische Friedrich-Wilhelms-Universitat, Bonn
  - DIAKO Ev. Diakonie Krankenhaus gGmbH, Bremen
  - Medizinische Klinik Am Lukas - Krankenhaus, Bünde
  - General Hospital, Celle
  - Hospital Kuchwald Chemnitz, Chemnitz
  - Praxis Fuer Haematologie Internistische Onkologie, Cologne
  - Medizinische Universitaetsklinik I at the University of Cologne, Cologne
  - Cologne-Kalk
  - Carl - Thiem - Klinkum Cottbus, Cottbus
  - Klinikum Darmstadt, Darmstadt
  - Saint Johannes Hospital Dortmund, Dortmund
  - Universitatsklinikum Carl Gustav Carus, Dresden
  - St. Johannes Hospital - Medical Klinik II, Duisburg
  - Franz Hospital Dulmen, Dülmen
  - Florence-Nightingale-Krankenhause, Deaconess Kaiserswerth, Düsseldorf
  - Hans - Susemihl - Krankenhaus, Emden
  - Klinikum Erfurt, Erfurt
  - St. Antonius Hospital, Eschweiler
  - Universitaetsklinikum Essen, Essen
  - Evangelisches Krankenhaus Essen-Werden, Essen
  - Krankenhaus Nordwest, Frankfurt
  - Klinikum Frankfurt (Oder) GmbH, Frankfurt (Oder)
  - Evang. Deaconess Hospital Freiburg, Freiburg im Breisgau
  - Municipal Hospital Complex, Fulda
  - Robert - Koch Hospital, Gehrden
  - Centre for Internal Medicine Gießen, Giessen
  - Universitaetsklinikum Göttingen, Göttingen
  - Klinik Fuer Innere Medizin, Hematology/Oncology, Ernst Moritz Armdt Universitaet, Greifswald
  - Staedtisches Klinikum Guetersloh, Gütersloh
  - St. Marien Hospital - Katholisches Krankenhaus Hagen gGmbH, Hagen
  - Allgemeines Krankenhaus Hagen, Hagen
  - Krankenhaus St. Elisabeth und St. Barbara, Halle
  - Krankenhaus Martha-Maria Halle-Doelau gGmbH, Halle
  - Universitaetsklinikum Halle, Halle
  - Hamburg
  - Universitaetsklinikum Hamburg-Eppendorf, Hamburg
  - Asklepios Klinik Nord Heidberg, Hamburg
  - Allgemeines Krankenhaus Altona, Hamburg
  - Haematologisch-Onkologische Praxis Altona, Hamburg
  - Evangelische Krankenhaus Hamm, Hamm
  - Hanover
  - Krankenhaus Siloah - Medizinische Klinik II, Hanover
  - Henriettenstiftung Krankenhaus, Hanover
  - Medizinische Hochschule Hannover, Hanover
  - Oncology Specialists Clinic, Harrislee
  - Medizinische Universitaetsklinik und Poliklinik, Heidelberg
  - Thoraxklinik Heidelberg, Heidelberg
  - Regional Hospital Heidenheim, Heidenheim
  - Regional Hospital Am Plattenwald - Bad Friedrichhall, Heilbronn
  - Klinikum Herford, Herford
  - Marienhospital at Ruhr University Bochum, Herne
  - Privatklinik Dr. R. Schindlbeck GmbH & Co. KG, Herrsching am Ammersee
  - Onkologische Schwerpunktpraxis, Hildesheim
  - Evang. Hospital, Holzminden
  - Medical University Hospital Homburg, Homburg
  - Universitaetsklinikum des Saarlandes, Homburg
  - Hospital Complex Hoyerswerda, Hoyerswerda
  - Gemeinschaftspraxis Innere Medizin, Jena
  - Klinikum der Friedrich-Schiller Universitaet Jena, Jena
  - Municipal Hospital Complex of the University, Kaiserslautern
  - Staedtisches Klinikum Karlsruhe gGmbH, Karlsruhe
  - Red Cross Hospital Kassel, Kassel
  - Staedtisches Krankenhaus Kiel, Kiel
  - Praxis fuer Haematologie und Onkologie, Koblenz
  - Stiftungsklinikum Mittelrhein - Gesundheitszentrum Evangelisches Stift Sankt Martin Koblenz gGmbH, Koblenz
  - Kliniken der Stadt Koeln gGmbH - Krankenhaus Merheim, Koln-Merheim
  - Leonardis Clinic, Kornwestheim
  - Klinikum Krefeld GmbH, Krefeld
  - Frankenwald Klinik, Kronach
  - Caritas - Krakenhaus Lebach, Lebach
  - Medizinische Klinik und Poliklinik III - Universitaetsklinikum Leipzig, Leipzig
  - University Leipzig Clinic of Internal Medicine, Leipzig
  - Leipzig
  - Staedtisches Klinikum "St. Georg" Leipzig, Leipzig
  - Klinikum Lippe - Lemgo, Lemgo
  - St. Vincenz Hospital Limburg, Limburg
  - St. Bonifatius Hospital Lingen, Lingen
  - Dreifaltigkeits Hospital, Lippstadt
  - Klinikum Ludwigsburg, Ludwigsburg
  - Klinikum der Stadt Ludwigshafen am Rhein, Ludwigshafen
  - St. Marien Hospital Ludwighafen, Ludwigshafen
  - Universitaetsklinikum Schleswig-Holstein - Campus Luebeck, Lübeck
  - Staedtisches Klinikum Magdeburg - Altstadt, Magdeburg
  - Universitaetsklinkum Magdeburg der Otto-von-Guericke-Universitaet Magdeburg, Magdeburg
  - Johannes Gutenberg University, Mainz
  - German CML Study Group, Manheim
  - Marburg
  - Philipps-Universitaet Marburg Klinikum, Marburg
  - Regional Hospital Mayen, Mayen
  - Klinikum Minden, Minden
  - Minden
  - Ev. Hospital Bethesda, Monchenglabach
  - Monchenglasbach/Rheydt
  - Hospital Maria-Hilf II, Mönchengladbach
  - Krankenhaus Muenchen Schwabing, Munich
  - Klinikum der Universitaet Muenchen - Grosshadern Campus, Munich
  - Evangelisches Krankenhaus - Mülheim, Mülheim
  - St. Marien Hospital - Muelheim an der Ruhr, Mülheim
  - Kreiskrankenhaus Muenchberg, Münchberg
  - Munich Oncologic Practice at Elisenhof, München
  - Klinikum der Universitaet Muenchen - Innenstadt Campus, München
  - Medizinische Klinik und Poliklinik A - Universitaetsklinikum Muenster, Münster
  - Regional Hospital Neumarkt, Neumarkt
  - Staedtisches Klinikum Neunkirchen gGmbH, Neunkirchen
  - Lukaskrankenhaus Neuss, Neuss
  - Klinikum Nuernberg - Klinikum Nord, Nuremberg
  - Klinikum Offenburg, Offenburg
  - Hematologische Praxis, Oldenburg
  - Ev. Hospital Oldenburg, Oldenburg
  - Klinikum Oldenburg, Oldenburg
  - Paracelsus - Klinik Osnabrück, Osnabrück
  - Municipal Hospital Complex, Pforzheim
  - Klinikum Ernst Von Bergmann, Potsdam
  - Kreiskrankenhaus Radebeul, Radebeul
  - Krankenhaus St. Elisabeth - Ravensburg, Ravensburg
  - Klinikum der Universitaet Regensburg, Regensburg
  - Hematologische Onkologische Praxis, Regensburg
  - Krankenhaus Barmherzige Brueder Regensburg, Regensburg
  - Jakobi Krankenhaus, Rheine
  - Klinik und Poliklinik fuer Innere Medizin - Universitaet Rostock, Rostock
  - Klinik und Poliklinik fuer Strahlentherapie - Universitaetsklinikum Rostock, Rostock
  - Rostock
  - Caritasklinik St. Theresia, Saarbrücken
  - Schwerpunktpraxis fuer Haematologie und Onkologie, Saarbrücken
  - St. Elizabeth-Klinik Saarlouis, Saarlouis
  - Martin - Luther Hospital, Schleswig
  - Deaconess Hospital, Schwäbisch Hall
  - Leopoldina - Krankenhaus, Schweinfurt
  - Evang. Jung-Stilling Hospital, Siegen
  - St. Lukas - Clinic Solingen, Solingen
  - Klinik fuer Onkologie - Katharinenhospital Stuttgart, Stuttgart
  - Diakonie Klinikum Stuttgart, Stuttgart
  - Klinikum Stuttgart - Buergerhospital, Stuttgart
  - Hospital Bad Cannstatt, Stuttgart
  - Robert-Bosch-Krankenhaus, Stuttgart
  - St. Elisabeth Hospital Thuine, Thuine
  - Regional Hospital Traunstein, Traunstein
  - Krankenanstalt Mutterhaus der Borromaerinnen, Trier
  - Trier
  - Krankenhaus Der Barmherzigen Brueder, Trier
  - Hospital Tutzing, Tutzing
  - Comprehensive Cancer Center Ulm at Universitaetsklinikum Ulm, Ulm
  - Ev. Hospital Unna, Unna
  - St. Marienhospital - Vechta, Vechta
  - Klinikum Der Stadt Villingen - Schwenningen, Villingen-Schwenningen
  - Regional Hospital Waldbrol, Waldbröl
  - Hospital Wetzler, Wetzlar
  - Deutsche Klinik fuer Diagnostik, Wiesbaden
  - Dr. Horst-Schmidt-Kliniken, Wiesbaden
  - Ev. Hospital Witten-Herdecke, Witten
  - Kliniken St. Antonius, Wuppertal
  - University Wurzburg, Würzburg
  - Municipal Hospital Complex Zwickau, Zwickau
- Switzerland (2):
  - UniversitaetsSpital Zuerich, Zurich
  - City Hospital Triemli, Zurich

REFERENCES:
- [Background] Trumper L, Zwick C, Ziepert M, Hohloch K, Schmits R, Mohren M, Liersch R, Bentz M, Graeven U, Wruck U, Hoffmann M, Metzner B, Hasenclever D, Loeffler M, Pfreundschuh M; German High-Grade Non-Hodgkin's Lymphoma Study Group (DSHNHL). Dose-escalated CHOEP for the treatment of young patients with aggressive non-Hodgkin's lymphoma: I. A randomized dose escalation and feasibility study with bi- and tri-weekly regimens. Ann Oncol. 2008 Mar;19(3):538-44. doi: 10.1093/annonc/mdm497. Epub 2008 Jan 22. PMID 18212092
- [Result] Pfreundschuh M, Zwick C, Zeynalova S, Duhrsen U, Pfluger KH, Vrieling T, Mesters R, Mergenthaler HG, Einsele H, Bentz M, Lengfelder E, Trumper L, Rube C, Schmitz N, Loeffler M; German High-Grade Non-Hodgkin's Lymphoma Study Group (DSHNHL). Dose-escalated CHOEP for the treatment of young patients with aggressive non-Hodgkin's lymphoma: II. Results of the randomized high-CHOEP trial of the German High-Grade Non-Hodgkin's Lymphoma Study Group (DSHNHL). Ann Oncol. 2008 Mar;19(3):545-52. doi: 10.1093/annonc/mdm514. Epub 2007 Dec 6. PMID 18065407